CLINICAL TRIAL: NCT02029885
Title: Wave IV Study: Phase II Randomized Sham Controlled Study of Renal Denervation for Subjects With Uncontrolled Hypertension
Brief Title: Sham Controlled Study of Renal Denervation for Subjects With Uncontrolled Hypertension
Acronym: WAVE_IV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kona Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KM14-001
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Hypertension
Keywords: Hypertension; Renal Denervation
MeSH Terms: conditions — Hypertension | interventions — Therapies, Investigational

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Investigational Therapy (Surround Sound) (Experimental): Investigational Therapy using external focused ultrasound
  Interventions: Device: Investigational Therapy (Surround Sound)
- Sham Control (Sham Comparator): Blinded Sham Control Arm
  Interventions: Device: Sham Control

INTERVENTIONS:
Device: Investigational Therapy (Surround Sound)
  Arms: Investigational Therapy (Surround Sound)
Device: Sham Control
  Arms: Sham Control

SUMMARY:
To demonstrate that non-invasive renal denervation is safe and shows a net difference in blood pressure reduction when compared to sham in subjects with uncontrolled hypertension.

DETAILED DESCRIPTION:
This study is a sham controlled, double blind study of subjects with uncontrolled hypertension consisting of two arms, sham and therapy. Bilateral renal denervation will be performed non-invasively using the Kona Medical Surround Sound System which delivers focused ultrasound therapy to ablate the nerves surrounding the renal artery utilizing real time ultrasound for targeting and tracking.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age and no more than 90 years of age
2. Average SBP ≥ 160 mmHg
3. 24 hour average ABPM daytime SBP ≥ 135 mmHg.
4. No medication changes for a minimum of 1 months prior to screening.
5. At minimum, subject must be on at least three antihypertensive medications, with one being a diuretic, and each must meet one or more of the following full dose criteria:

   1. Highest labeled dose according to medication's labeling;
   2. Highest usual dose per clinical guidelines JNC-7;
   3. Highest tolerated dose; and/or
   4. Highest appropriate dose for the subject per the PI's clinical judgment.
6. Subject has two functioning kidneys.
7. Subject has an eGFR value of ≥ 30 ml/min/1.73 m² (MDRD formula).

Exclusion Criteria:

1. Subject has any secondary cause of hypertension
2. Subject has evidence of clinically significant renal artery stenosis as determined by flow rate, velocity and Doppler analysis on ultrasound
3. Subject has kidney stones that are of a size and location that are determined at discretion of the investigator to potentially interfere with treatment
4. Subject has a history of intra-abdominal surgery within the past six months
5. Subject has heterogeneities in the kidney such as large cysts or tumors that are determined at discretion of the investigator to potentially interfere with treatment.
6. Stenotic valvular heart disease for which BP reduction would be hazardous as determined by referring physician.
7. MI, unstable angina, or CVA in the prior 6 months.
8. Known severe primary pulmonary HTN
9. Subject has a history of myocardial infarction, unstable angina pectoris, or cerebrovascular accident within the last six months.
10. Subject has hemodynamically significant valvular heart disease.
11. Subject has BMI over 40 km/m^2
12. Subject has a target treatment depth over 13 cm.
13. Subject has anatomy that precludes treatment with the Kona Medical Surround Sound System.
14. Subject is pregnant, nursing, or intends to become pregnant during the trial period.
15. Subject is currently enrolled in other potentially confounding research.
16. Subject has any condition that, at the discretion of the investigator, would preclude participation in the trial.
17. Subject is unable, or unwilling, to comply with the protocol-required follow-up schedule

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Safety at 6 weeks follow-up | 6 weeks
  Safety will be assessed by incidence of Major Adverse Events (MAE), defined as a composite of the following events at 6-weeks follow-up.
  * All cause mortality;
  * End-stage Renal Disease defined as eGFR < 15 ml/min or need for renal replacement therapy
  * Hospitalization for hypertensive crisis not related to confirmed non-adherence with medications as assessed by toxicological and other medical analyses and testing.
  OR
  - New renal artery stenosis > 70% confirmed by angiography within 6 months of randomization
Change in OBP | 6 months
  Change in Office Systolic Blood Pressure (OBP) as measured from screening visit one to the 6 month post randomization follow-up visit.

SECONDARY OUTCOMES:
Change in ABPM | 6 months
  Change in average 24-hour ambulatory blood pressure from screening to the 6 month follow-up visit

OTHER OUTCOMES:
Chronic Safety | 6 months
  Chronic safety is assessed and compared between the control and treatment groups at 6 months post-randomization as follows:
  * Cardiovascular/Renal Death;
  * End stage Renal Disease
  * Increase in serum creatinine of > 50%; and
  * Hospitalization for hypertensive crisis not confirmed non-adherence with medications.
Reduction in blood pressure | 6 months
  Reduction in systolic and diastolic blood pressure as compared between groups at time points through the 6 month follow-up period for interval differences of 10,15 and 20 mmHg.
Incidence of achieving target OBP | 6 months
  Incidence of achieving target OBP (< 140 mmHg) through the 6 month follow-up period.
Reduction in anti-hypertensive medications | 6 months
  Incidence of reductions in the number of anti-hypertensive medications and reductions in the doses of anti-hypertensive medications.
Changes in OBP | 24 months
  Changes in OBP from screening to the 12, 18, and 24 month follow-up periods.
Changes in HR | 6 months
  Changes in HR (as measured by OBP and ABPM) through the 6 month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Schmieder, MD, Principal Investigator — University Hospital of University of Erlangen-Nuremberg
Locations (28):
- Monash Medical Centre, Clayton, Australia
- Medizinischen Universität Wien -UK für Klinische Pharmakologie, Vienna, Austria
- Colombia (2):
  - Angiografia de Occidente, S.A., Cali
  - CHD Cardio Centro de Excelencia SAS, Cali
- Czechia (5):
  - St. Anne's University Hospital, Brno
  - University Hospital Brno, Brno
  - Městská Nomocnice Ostrava, Ostrava
  - General University Hospital, Prague
  - Nemocnice Na Homolee Hospital, Prague
- Germany (9):
  - University Hospital Bonn, Bonn
  - Uniklinik Köln, Cologne
  - University Hospital of the University of Erlangen-Nuremberg, Erlangen
  - CardioVascular Center Frankfurt - Sankt Katharinen Hospital, Frankfurt
  - University Hospital Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Leipzig, Leipzig
  - Sana CardioMed Nord, Lübeck
  - Deutsches Herzzentrum Muenchen, Munich
  - Clemens Hospital GmbH, Münster
- Mercy Angiography, Aukland, New Zealand
- Poland (2):
  - Oddział Kliniczny II Kliniki Kardiologii, Krakow
  - Institute Of Cardiology, Warsaw
- United Kingdom (7):
  - Birmingham Heartlands Hospital, Birmingham
  - University Hospital Wales, Cardiff
  - Royal Devon and Exeter Hospital, Exeter
  - University of Glasgow, Glasgow
  - St. Bartholomew's Hospital, London
  - University College London, London
  - Southampton University Hospital, Southampton

REFERENCES:
- [Derived] Saxena M, Shour T, Shah M, Wolff CB, Julu POO, Kapil V, Collier DJ, Ng FL, Gupta A, Balawon A, Pheby J, Zak A, Rull G, O'Brien B, Schmieder RE, Lobo MD. Attenuation of Splanchnic Autotransfusion Following Noninvasive Ultrasound Renal Denervation: A Novel Marker of Procedural Success. J Am Heart Assoc. 2018 Jun 12;7(12):e009151. doi: 10.1161/JAHA.118.009151. PMID 29895590